CLINICAL TRIAL: NCT06337708
Title: Smart Walk: An Efficacy Trial of a Culturally Tailored Smartphone-Delivered Physical Activity Intervention for African American Women
Brief Title: Smart Walk: A Culturally Tailored Smartphone-Delivered Physical Activity Intervention for African American Women
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00017286; R01HL168170 (NIH)
Record Dates: First submitted 2024-01-29; First posted 2024-03-29 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Physical Activity; Exercise; Heart Diseases; Diabetes Mellitus; Physical Inactivity
Keywords: mHealth; women's health; health equity; African American women; Black women; exercise; physical activity; heart disease; diabetes
MeSH Terms: conditions — Motor Activity; Heart Diseases; Diabetes Mellitus; Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smart Walk (Experimental): Participants will receive a culturally tailored smartphone-delivered physical activity intervention.
  Interventions: Behavioral: Smart Walk
- Fitbit (Active Comparator): Participants will receive a Fitbit Inspire 3 activity monitor.
  Interventions: Behavioral: Fitbit

INTERVENTIONS:
Behavioral: Smart Walk — Smart Walk is a culturally tailored, Social Cognitive Theory-based multi-component smartphone delivered physical activity (PA) promotion intervention that delivered through the Smart Walk application, virtual physical activity coaching, and text messages. The Smart Walk smartphone application includes four key features: 1) personal profile pages, 2) culturally relevant multi-media physical activity promotion modules, 3) discussion boards, and 4) physical activity self-monitoring/tracking feature that integrates with Fitbit activity monitors for participants to track their daily, weekly, and monthly activity. Virtual physical activity coaches will actively engage and facilitate group-based dialogue among participants on the app discussion boards and provide individualized, one-on-one PA coaching via telephone or commercially available app-based video teleconferencing software (i.e., FaceTime, Zoom, Google hangouts).
  Arms: Smart Walk
Behavioral: Fitbit — This intervention group will receive a Fitbit activity monitor and be encouraged to use the commercially available device to increase physical activity.
  Arms: Fitbit

SUMMARY:
The purpose of this study is to test a culturally tailored, smartphone-delivered intervention designed to increase physical activity and reduce risk for heart disease and type 2 diabetes among African American women.

DETAILED DESCRIPTION:
This study addresses major public health concerns among African American women: physical inactivity and cardiometabolic disease risk.

African American women experience a high burden of cardiometabolic diseases, including heart disease, obesity, and type 2 diabetes. Regular aerobic physical activity is an established behavior to prevent and treat these conditions. Yet, the many African American women are insufficiently active, with only 27-40% meeting national aerobic physical activity guidelines.

This study will test the efficacy of Smart Walk, a culturally tailored, theory-based smartphone-delivered intervention designed to increase physical activity and improve cardiometabolic disease risk factors among African American women. In a 12-month trial, participants will be randomly assigned to either the Smart Walk intervention or a Fitbit-only comparison arm for an active 4-month intervention period, followed by an 8-month minimal contact follow-up period.

Specific Aims:

1. Test the effects of Smart Walk to increase physical activity and promote adherence to national aerobic physical activity guidelines; compared to Fitbit-only comparison group.
2. Test the effects of Smart Walk to improve cardiometabolic risk factors; compared to Fitbit-only comparison group.
3. Compare cost and cost effectiveness of the two intervention groups from a societal perspective.
4. Examine if protocol adherence predicts outcomes and potential mediation and moderation of intervention effects on physical activity and cardiometabolic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported African American/Black female
* Aged of 24-65 years
* Insufficiently Active (< 60 minutes of moderate-to-vigorous physical activity per week as measured by Exercise Vital Sign Questionnaire)
* BMI > 30 kg/m2
* English speaking and reading
* Ownership of a smartphone with the ability to download applications (i.e., apps)
* Ownership of a smartphone with the ability to receive text messages
* Willingness to receive a physical activity intervention delivered through their smartphone
* Willingness to include their first name or create an alias to be used on their profile page on the Smart Walk app

Exclusion Criteria:

* Plans to relocate out of Phoenix area in next 12 months
* Endorsing an item on the Physical Activity Readiness Questionnaire (PAR-Q), unless a doctor's note for study participation in provided
* Resting systolic blood pressure greater than 180 mmHG and/or a diastolic blood pressure greater than 120 mmHG , as assessed at baseline or at any other study assessment
* Self-reported participation in another diet or weight loss study at screening
* Pregnant or planning to become pregnant in the next 12 months

Ages: 24 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in accelerometer-measured moderate-to-vigorous intensity physical activity from baseline to 4- and 12-months | Assessed at baseline, 4-months, 12-months
  Participants will wear wrist-worn ActiGraph GT9X Link Activity monitors the activity monitor on their non-dominant wrist during all waking hours for 7 consecutive days to provide an assessment of usual activity
Change in self-reported moderate-to-vigorous intensity physical activity from baseline to 4- and 12-months | Assessed at baseline, 4-months, 12-months
  Assessed by the 7-Day Physical Activity Recall

SECONDARY OUTCOMES:
Change in cardiorespiratory fitness from baseline to 4- and 12-months | Assessed at baseline, 4-months, 12-months
  A modified Balke treadmill protocol will be used to estimate maximal aerobic capacity (i.e., VO2 peak).
Change in aortic pulse wave velocity from baseline to 4- and 12-months | Assessed at baseline, 4-months, 12-months
  A measure of aortic stiffness and will be assessed using SphygmoCor XCEL system using validated methodology.
Change in body weight from baseline to 4- and 12-months. | Assessed at baseline, 4-months, 12-months
  Measured in kilograms using an electronic scale
Change in body mass index from baseline to 4- and 12-months | Assessed at baseline, 4-months, 12-months
  Calculated using the formula: weight (in kilograms) / height (in meters)squared
Change in waste circumference from baseline to 4- and 12-months | Assessed at baseline, 4-months, 12-months
  Measured in centimeters
Change in blood pressure (mmHG) from baseline to 4- and 12-months | Assessed at baseline, 4-months, 12-months
  Both systolic and diastolic blood pressure will be assessed using electronic sphygmomanometer following 5-min rest
Change in tumor necrosis factor-alpha (TNF-α) from baseline to 4- and 12-months | Assessed at baseline, 4-months, 12-months
  Measured in serum using a commercial multiplex immunoassay platform; blood will be drawn after a 10 hour fast.
Change in interleukin 6 (IL-6) from baseline to 4- and 12-months | Assessed at baseline, 4-months, 12-months
  Measured in serum using a commercial multiplex immunoassay platform; blood will be drawn after a 10 hour fast.
Change in interleukin 10 (IL-10) from baseline to 4- and 12-months | Assessed at baseline, 4-months, 12-months
  Measured in serum using a commercial multiplex immunoassay platform; blood will be drawn after a 10 hour fast.
Change in interleukin 15 (IL-15) from baseline to 4- and 12-months | Assessed at baseline, 4-months, 12-months
  Measured in serum using a commercial multiplex immunoassay platform; blood will be drawn after a 10 hour fast.
Change in fasting blood glucose glucose from baseline to 4- and 12-months | Assessed at baseline, 4-months, 12-months
  Plasma glucose assessed after a 10 hour fasting blood draw. Measured using an automated chemistry analyzer.
Change in serum insulin from baseline to 4- and 12-months | Assessed at baseline, 4-months, 12-months
  Serum insulin collected after a 10 hour fasting blood draw.
Change in serum lipids (mg/DL) from baseline to 4- and 12-months | Assessed at baseline, 4-months, 12-months
  Triglycerides, total cholesterol, LDL-C, and HDL-C will be assessed
Change in insulin sensitivity (µIU/mL) from baseline to 4- and 12-months | Assessed at baseline, 4-months, 12-months
  Assessed by calculating homeostatic model assessment (HOMA) scores as: glucose (mg/dl) x insulin (μU/ml)/405.
Change in exercise self-efficacy from baseline to 4- and 12-months | Assessed at baseline, 4-months, 12-months
  Assessed by the 12-item Exercise Self-Efficacy survey (Sallis et al.1987). The range of possible scores for this measure is 1-5, with higher scores indicating higher levels of physical activity self-efficacy.
Change in self-regulation for physical activity from baseline to 4- and 12-months | Assessed at baseline, 4-months, 12-months
  Assessed by the 10- item Self-Regulation Scale from the Health Beliefs Survey (Anderson-Bill 2006). This scale assesses the use of behavioral strategies to incorporate physical activity into daily activities (i.e., take stairs instead of elevator, walking instead of driving when running errands). The range of possible scores for this measure is 1-5, with higher scores indicating higher levels of physical activity self-regulation.
Change in social support for physical activity from baseline to 4- and 12-months | Assessed at baseline, 4-months, 12-months
  Assessed by the Social Support for Exercise survey developed by Sallis et al (1987). This scale assesses social support from family support (10-items, with a possible range of scores from 10-50) and friends (8-items, with a possible score range from from 8-40). Higher scores indicate greater levels of social support.
Change in outcome expectations for physical activity from baseline to 4- and 12-months | Assessed at baseline, 4-months, 12-months
  Assessed using the 9-item Outcome Expectation Scale for Exercise scale, developed by Resnick (2000). The range of possible scores for this measure is 1-5, with higher scores indicating more positive expectancies associated with physical activity engagement.
Change in behavioral capability for physical activity from baseline to 4- and 12-months | Assessed at baseline, 4-months, 12-months
  Assessed using a 6-item scale developed by the research team in previous research. The range of possible scores for this measure is 1-6, with higher scores indicating higher levels of behavioral capability of physical activity.

OTHER OUTCOMES:
Treatment acceptance | Assessed at 4-months and 12-months
  Survey assessing acceptance, feasibility, and consumer satisfaction of intervention.
Protocol Adherence | Assessed at 4-months and 12-months
  Fitbit wear, app utilization, and adherence to physical activity coaching session protocols will be assessed as moderators.
Program costs | Assessed at 4-months and 12-months
  Costs borne by the program, including Fitbit activity monitors, Smart Walk app development, and all personnel salaries/hourly wages.
Participant costs | Assessed at 4-months and 12-months
  Participant costs associated with study participation, including time spent using the Smart Walk app, time spent in physical activity coaching, and cellular phone data charges over their plan limit.
Cost-effectiveness | Assessed at 4-months and 12-month
  Cost effectiveness will be evaluated by combining the mean total cost per participant with effectiveness (baseline to 12-month changes in minutes/week of moderate-to-vigorous physical activity). We will calculate the incremental cost effectiveness ratios (ICER) for the Smart Walk intervention compared to the Fitbit comparison arm.
Objectively-measured home neighborhood characteristics | Assessed at baseline
  GIS mapping and computer vision techniques will be used to assess macro-scale and micro-scale home neighborhood environment characteristics of participants.
Subjectively-measured Neighborhood environment walkability | Assessed at baseline
  Subjectively-measured Neighborhood Environment Walkability will be measured using the Neighborhood Environment Walkability Scale (NEWS). This measure includes 43 items and assesses the following environmental characteristics: residential density (6-items, possible range of scores range 1-5), land use mix-diversity (22 items, possible range of scores range 1-5), street connectivity (2 items, possible range of scores range 1-4), walking/cycling facilities (6 items, possible range of scores range 1-4), aesthetics (4 items, possible range of scores 1-4), pedestrian/traffic safety (3 items, possible range of scores 1-4). Higher scores indicate greater walkability.
Race-related Stress | Assessed at baseline
  Race-related stress, as a result of experiencing individual, cultural and institutional racism, will be assessed using the 22-item Index of Race-Related Stress-Brief survey. This survey has a possible score range of 0 to 88, with higher scored indicating greater stress as a result of experiencing racism.
Perceived Structural Racism | Assessed at baseline
  Structural racism will be assessed using the 20-item Perceived Structural Racism Scale. This scale has a possible scoring range of 20-120 with higher scores indicating greater levels of perceived structural racism.

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided